CLINICAL TRIAL: NCT06069310
Title: Evaluation of Mepolizumab Effectiveness in Patients With Chronic Rhinosinusitis With Nasal Polyps and Comorbid Severe Eosinophilic Asthma: an Integrative Multi-omics Approach to Assess Biomarker Signatures of Responsive Disease Endotypes
Brief Title: Mepolizumab Effectiveness in Patients With Chronic Rhinosinusitis, Nasal Polyps and Comorbid Severe Eosinophilic Asthma
Acronym: MepoRiNaPAs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Paraskevi Katsaounou, Associate Professor of Respiratory Medicine, National and Kapodistrian University of Athens
Other Study IDs: 14919
Record Dates: First submitted 2023-09-06; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Severe Eosinophilic Asthma; Chronic Rhinosinusitis Without Nasal Polyps
Keywords: Chronic Rhinosinusitis; Severe Eosinophilic Asthma; Microbiome; Nasal Polyps; Mepolizumab
MeSH Terms: conditions — Pulmonary Eosinophilia; Nasal Polyps | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum blood and nasal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control subjects: Healthy control subjects withouth asthma nor chronic rhinosinusitis or other chronic respiratory diseases
- Chronic rhinosinusitis with nasal polyps (CRSwNP) patients with comorbid severe asthma: Patients that have chronic rhinosinusitis with nasal polyps (CRSwNP) and comorbid severe asthma will be enrolled
  Interventions: Drug: Mepolizumab 100 MG
- Chronic rhinosinusitis with nasal polyps (CRSwNP) patients without asthma: Patients that have chronic rhinosinusitis with nasal polyps (CRSwNP) without asthma will be enrolled
  Interventions: Drug: Mepolizumab 100 MG

INTERVENTIONS:
Drug: Mepolizumab 100 MG — Monthly administartion of mepolizumab 100mg
  Other Names: nucala
  Groups: Chronic rhinosinusitis with nasal polyps (CRSwNP) patients with comorbid severe asthma; Chronic rhinosinusitis with nasal polyps (CRSwNP) patients without asthma

SUMMARY:
The goal of this observational study is to learn about clinical and functional outcomes in patients with Chronic rhinosinusitis with nasal polyps and comorbid Severe Eosinophilic Asthma and patients with Chronic rhinosinusitis with nasal polyps only treated with mepolizumab compared to healthy controls.

Participants will be asked to give nasal, blood and sputum samples before mepolizumab administration (T0) and at 3 (T3), 6 (T6) and 12 (T12) months after mepolizumab initiation The main aims are to identify airways microbiota modifications and differential gene expression after mepolizumab initiation.

Researchers will compare:

* Patients with Chronic rhinosinusitis with nasal polyps and comorbid Severe Eosinophilic Asthma
* Patients with Chronic rhinosinusitis with nasal polyps only
* Healthy subjects

The research will address the following questions:

1. What are the prospective clinical and functional outcomes of mepolizumab treatment
2. What is the impact of mepolizumab therapy on the airways microbiota and how this may relate to a potentially reduced need for steroids
3. What are the host differential gene expression patterns and the immune/inflammatory (cytokines/chemokines) profile alterations in airways microenvironment and in systemic circulation in response to therapy
4. What are the associations between host and microbiome variables for building up diagnostic and predictive biomarker classifiers of responsive disease endotypes

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) has been divided into two subtypes: CRS with (CRSwNP) and without nasal polyps (CRSsNP), which not only differ in terms of presence of polyps, but also appear to have distinct pathogenesis and clinical presentations. It is known that CRSwNP patients have a greater disease burden compared with those suffering from CRSsNP with respect to disease severity and poor treatment. More specifically, approximately 85% of CRSwNP patients are characterized by severe symptoms, recurrent disease and a dominant Th2 endotype associated with a marked infiltration of eosinophils and mast cells, goblet hyperplasia and increased levels of Th2 inflammatory cytokines including Interleukin IL-4, IL-5, and IL-13. An additional hallmark of CRSwNP is the loss of healthy barrier function in sinonasal epithelial cells, increased permeability, decreased epithelial resistance, and a high degree of tissue remodeling compared with cells from CRSsNP patients and control individuals. This loss of barrier function is reflective of a general inflammatory process, though it is unclear if the epithelial cells are inherently abnormal or if the state is induced. Treatment for CRS is most frequently glucocorticoid-based, but response is quite variable in patients with nasal polyps and side-effects from oral steroids limit their long-term efficacy. An inverse relationship between glucocorticoid receptor β expression in nasal polyp tissue and steroid efficacy has been observed. Furthermore, neutrophil accumulation in nasal polyp tissue has been related to corticosteroid insensitivity. Some individuals exhibit a very high level of resistance to steroid therapy thus underscoring the need for therapeutics targeting non-steroid-responsive pathophysiologic mechanisms involved in sinus polyp formation.

Asthma is frequently a comorbid condition sharing similar pathophysiology in CRSwNP patients, which affects 20-60% of diseased individuals. Yet, specific subsets of patients such as those with IL-5-enriched nasal polyps are characterized by a greater percentage of asthma and revision surgery. Clinically, CRSwNP with comorbid asthma (CRSwNP + AS) is associated with even more severe sinonasal symptoms and worse quality of life, and it is more difficult to treat both medically and surgically. Correspondingly, asthma in the presence of nasal polyposis is harder to control, being more exacerbation prone, with increased airway obstruction and more extensive eosinophilic inflammation.

Although a clear correlation apparently exists between sinonasal and lower airway inflammation in patients with CRSwNP+AS, the definitive underlying mechanism(s) remains poorly elucidated. The airways microbiota, i.e. the niche-specific communities of microbes including bacteria, fungi, archaea and viruses that inhabit the respiratory tract, has been proved to play a critical role in airway health and immune cells homeostasis -including eosinophils regulation- through its constant interaction with the mucosal immune system. Alterations in the composition and diversity of microbiome across the respiratory tract may contribute to the observed inflammatory crosstalk in CRSwNP + AS, and perhaps influence patients' response to treatment. Nasal and lower airway microbiota dysbiosis have been proved to be implicated in the persistence of characteristic inflammatory endotypes in both CRSwNP and asthma. It has been shown that bacterial dysbiosis is correlated with CRS status and that specific microbiota taxonomic classifications are correlated with patient phenotypes, including the presence of nasal polyps. A high proportion of patients with CRSwNP are colonized with Staphylococcus (S.) aureus and IgE antibodies to S. aureus enterotoxins are frequently found in diseased tissue specimens. Both S. aureus and Pseudomonas aeruginosa bacteria can disrupt the epithelial barrier contributing to presumed physiologic mechanisms for CRSwNP development. It has been previously demonstrated that S. aureus is able to drive Th2 type inflammation in CRSwNPand that the expression of IL-5 and of IgE against S. aureus superantigens (SE-IgE) within polyp tissue is associated with comorbid asthma and CRSwNP recurrence. Furthermore, antimicrobial compounds including lysozyme, S100 proteins, and β-defensins all are decreased in CRSwNP patients compared to matched controls. This reduction in natural defenses could play a key role in shifting the balance towards dysbiosis. Furthermore, in addition to bacterial microbiome which has been the focus of most recent studies, the contribution of fungal microbiota to allergic airway diseases has been recently emerged. An alternative proposed pathogenic mechanism for Th2-biased CRS is that T-cells are allergically sensitized to fungi in the ambient environment, leading to allergic inflammation characterized by a Th2-high state. Overall, a distinct microbiome role in CRSwNP and asthma pathogenesis is actually recognized. However, the significance of interactions between the lower/upper airways flora and the host local and systemic inflammatory response has not yet been well defined neither such a knowledge is exploited for a more accurate patients classification and selection of best possible therapeutic manipulation to change disease progression.

Evidently, an optimal diagnostic approach for CRSwNP + AS would include use of very specific biomarkers ensuring a detailed endotyping, whereas, there is a growing consensus that both diseases should be treated to improve therapeutic outcome. However, the management of CRSwNP + AS patients who remain uncontrolled despite medical and often surgical intervention poses a great challenge to clinicians. Fortunately, there has been significant innovation and expansion in the treatment armamentarium since the advent of biological therapies. Targeted biologics (monoclonal antibodies against IL-4, IL-5, IL-13 and IgE) for treating asthma are now being used for CRSwNP with encouraging results.

Recently, mepolizumab (Nucala; GlaxoSmithKline), an anti-IL5 humanized mab known to efficiently down-regulate the eosinophilic inflammatory pathway and to exhibit clinical benefit in patients with severe, eosinophilic asthma, has completed a phase 3 trial (SYNAPSE; NCT03085797) including 413 subjects with CRSwNP. Early results showed treatment with mepolizumab had a significant difference in median nasal polyp score compared to baseline (-0.73; 95% CI: -1.11 to -0.34) and nasal obstruction visual analog score compared to baseline (-3.14; 95% CI: -4.09 to -2.18; unpublished data). However, there are only limited longitudinal studies evaluating this biologic's efficacy in CRSwNP+AS patients, while the assessment of action mode and biomarkers predicting responsiveness, remain to be elucidated.

Despite the persuasive rationale for systemic targeting of shared pathways in CRSwNP+AS with novel biologics, in clinical practice the nose and lungs are often treated as separate entities and these therapeutics are considered rather challenging for the clinicians due to their high cost and necessity for careful selection of patients and right treatment. Furthermore therapeutic decision-making is still based on a rather trial-and-error approach, resulting in treatment failures or relapses. There is clearly a need for a personalized medicine approach that would allow for a more accurate prediction of the appropriate choice of the drug at the initial assessment, and ideally would communicate chances of long-term success to an individual patient.

The principal goal of this three arms RWE study (CRSwNP+AS, CRSwNP-AS, healthy controls) study is to develop signatures of host-microbiome biomarkers of both diagnostic and predicting value in order to provide a rational guideline for mepolizumab selection in precision treatment of patients with CRSwNP+AS.

In this frame, mepolizumab therapeutic potential will be assessed in relation to the rather heterogeneous presentations of Th2 inflammation and airways microbiome structure. The protocol will take on the question of microbiome dysbiosis involvement in immune activation and dysfunction contributing to CRSwNP + AS diversity and delving into the complex patterns of host-microbiota molecular interactions in the upper and lower airways that may shape patients' clinical predisposition to mepolizumab therapy.

To address the study objectives a longitudinal design is proposed combining clinical assessments with high-throughput multi-omics analyses of patients' samples and advanced bioinformatics for data integration. The starting point of the project will be the consent recruitment of healthy controls, CRSwNP + AS and CRSwNP - AS participants. Collection of biological samples from patients and clinical assessment/measurements of cell counts will take place at baseline, i.e. the day of treatment initiation before mepolizumab administration (T0) and at 3 (T3), 6 (T6) and 12 (T12) months after mepolizumab initiation. Samples from healthy participants will be collected only at baseline (T0) and analyzed in parallel with the corresponding samples from CRSwNP patients. DNA and RNA will be isolated from induced sputum and nasal samples collected at T0 and T3 for subsequent 16S rRNA gene amplicon sequencing, DNA shot-gun sequencing (applied only in selected number of patients and healthy controls) and bulk RNA sequencing (RNAseq), to identify airways microbiota modifications and differential gene expression, respectively. Peripheral blood mononuclear cells (PBMC) from a representative number of patients and healthy controls will be also analyzed at the same time points by single-cell RNA sequencing (scRNAseq). In parallel, the dynamic pattern of cytokines/chemokines in serum/airways samples will be determined by xMAP immunoassays at T0 and T3. Subsequently, multiple comparisons at the level of microbiome and host parameters will be undertaken mainly through two paths. First, between patients and healthy controls at T0 to assess differences of disease versus "normal" condition; Second, pairwise in each patient at T0 and at time intervals, mostly at T3, after treatment intervention, to capture potential alterations in response to mepolizumab. Next, a thorough integrative analysis engaging clinical data and multi-omics data (from microbiome, bulk RNAseq, scRNAseq as well as cytokinome/chemokinome analyses) will be undertaken to investigate possible microbiome-host interactions. Finally, this integrative analysis will be exploited to gain a global view of hub genes, inflammatory mediators and microbial taxa involved in key interactions and to build biomarker signatures that might serve as indicators of specific disease subtypes and/or predictors of mepolizumab treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for inclusion will be patients diagnosed with CRSwNP according to the European Position Paper on Rhinosinusitis and Nasal Polyps that fulfill the criteria for initiating treatment with biologics as standard of care [49], suffering or not from comorbid severe asthma (CRSwNP + AS, CRSwNP - AS, respectively) who will consent to participate in the study. The study will not influence prescribing of mepolizumab to patients.

Eligible to treatment women in childbearing potential will be informed before consent that they must take care of contraception and potential pregnancy during therapy as there is not enough data regarding the use of mepolizumab during pregnancy. All patients with severe asthma will be qualified for treatment with mepolizumab in accordance with GINA guidelines.

Exclusion Criteria:

* Patients less than 18 years of age, subjects suffering from COPD, known or suspected immunodeficiency or autoimmune disease, chronic interstitial lung diseases, cystic fibrosis, individuals exposed to systemic corticosteroid/immunosuppressive treatments, biologics for asthma care or antibiotics within the previous 3 months before mepolizumab administration, active smokers and obese individuals will be excluded from this study. Pregnant women will not be included into the study because of the potential changes that their microbiome and other host parameters could undergo during pregnancy. The control group will comprise healthy volunteers who will be free from CRS, asthma, and atopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We estimate to recruit 40 CRSwNP patients (20 with and 20 without severe asthma) and 20 healthy control subjects. All participants will be adults (18 years and older) of both sexes. Clinical evaluation of CRSwNP and asthma will be made according to the European Position Paper on Rhinosinusitis and Nasal Polyps. Patients with significant sino-nasal disease and/or those who fail medical management will be evaluated for functional endoscopic sinus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Sino-nasal outcome test-22 (SNOT-22) score | at baseline and in 3, 6 and 12 months
  SNOT-22 score will be considered as a measure of post-treatment alterations in CRSwNP clinical symptoms
Asthma control test (ACT) | at baseline and in 3, 6 and 12 months
  ACT will assess potential treatment-induced alterations in asthma symptoms

SECONDARY OUTCOMES:
Mean change of nasal endoscopic polyps score | at baseline and in 3, 6 and 12 months
  Nasal endoscopic polyps score will be considered as a measure of post-treatment alterations in CRSwNP participants
Mean change of the polyposis severity visual analog scale (VAS) score | at baseline and in 3, 6 and 12 months
  Polyposis severity VAS score will estimate potential post-treatment changes in CRSwNP participants
Forced Expiratory Volume at 1 s % (%FEV1: FEV1/FEV1 predicted) and Morning Peak Expiratory Flow measurements | at baseline and in 3, 6 and 12 months
  FEV1: FEV1/FEV1 predicted and Morning Peak Expiratory Flow measurements will assess potential treatment-induced alterations in pulmonary function
Fractional Exhaled Nitric Oxide Testing (FENO) | at baseline and in 3, 6 and 12 months
  FENO measurements will assess potential treatment-induced alterations in airways inflamation
Forced oscillation technique (FOT) measurements at baseline and after 3, 6 and 12 months of mepolizumab treatment | at baseline and in 3, 6 and 12 months
  FOT measurements will estimate post-treatment changes in respiratory mechanics
Hospital Anxiety and Depression Scale (HADS) questionnaire | at baseline and in 3, 6 and 12 months
  HADS questionnaire will track evolution of psychological symptoms in response to treatment
Mean change from baseline in Asthma Quality of Life Questionnaire (AQLQ) | at baseline and in 3, 6 and 12 months
  AQLQA will assess changes in asthma-specific health-related quality of life in response to mepolizumab therapy
Mean change from baseline in immune cells (eosinophil/neutrophil) counts in nasal, sputum and blood samples | at baseline and in 3, 6 and 12 months
  Immune cells measurements will indicate the potential alterations in airway (nasal, sputum) and systemic (blood) inflammation in response to mepolizumab treatment
Mean change from baseline of cytokines/chemokines levels in blood and airways samples | at baseline and in 3 months
  Multiplex measurements of cytokines/chemokines levels will inform for treatment-induced alterations in airway (nasal, sputum) and systemic (blood) inflammation
Differential gene expression (fold changes) in nasal and sputum samples | at baseline and in 3 months
  Differential gene expression will evaluate the treatment-mediated alterations in the airway transcriptome
Differential single-cell gene expression (fold changes) of Peripheral Blood Mononuclear Cells (PBMC) from responders and non-responders to mepolizumab treatment | at baseline and in 3 months
  Differential single-cell gene expression analysis will estimate the potential treatment-induced changes in single-cell gene expression in responders versus non-responders to mepolizumab treatment
Mean change from baseline in airway (sputum, nasal) microbiome alpha and beta diversity indices at 3 months post-treatment in airway samples | at baseline and in 3 months
  Measurement of the alpha and beta microbiome diversity indices will assess the treatment-induced alterations in the microbiome characteristics
Differential abundances of microbial taxa (fold changes) from baseline at 3 months post-treatment in nasal and sputum samples | at baseline and in 3 months
  Differential taxa abundance will evaluate the treatment-mediated alterations in the abundance of specific airway microbial taxa
Differential abundances of predicted metabolic pathways (fold changes) from baseline at 3 months post-treatment in nasal and sputum microbiome | at baseline and in 3 months
  Differential abundance of metabolic pathways will estimate the treatment-mediated alterations in the microbiome function
Predictive biomarker classifiers of responsive disease endotypes | two years
  Harness associations between host and microbiome variables for building up diagnostic and predictive biomarker classifiers of responsive disease endotypes

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Katsaounou, MD, PhD, Msc, Principal Investigator — National Kapodistrian University of Athens; Eleni Loutrari, PhD, Study Director — National Kapodistrian University of Athens
Locations (2):
- Greece (2):
  - Pulmonary Dept First ICU, Evagelismos Hospital, Athens, Attica
  - Pulmonary Dept First ICU Evangelismos Hospital, Athens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banerji A, Piccirillo JF, Thawley SE, Levitt RG, Schechtman KB, Kramper MA, Hamilos DL. Chronic rhinosinusitis patients with polyps or polypoid mucosa have a greater burden of illness. Am J Rhinol. 2007 Jan-Feb;21(1):19-26. doi: 10.2500/ajr.2007.21.2979. PMID 17283555
- [Background] Kallieri M, Zervas E, Fouka E, Porpodis K, Mitrova MH, Tzortzaki E, Makris M, Ntakoula M, Papaioannou AI, Lyberopoulos P, Dimakou K, Koukidou S, Ampelioti S, Papaporfyriou A, Katsoulis K, Kipourou M, Rovina N, Antoniou K, Vittorakis S, Bakakos P, Steiropoulos P, Markopoulou K, Avarlis P, Papanikolaou IotaC, Markatos M, Gaki E, Samitas K, Glynos K, Papiris SA, Papakosta D, Tzanakis N, Gaga M, Kostikas K, Loukides S. RELIght: A two-year REal-LIfe study of mepolizumab in patients with severe eosinophilic asTHma in Greece: Evaluating the multiple components of response. Allergy. 2022 Sep;77(9):2848-2852. doi: 10.1111/all.15382. Epub 2022 May 30. No abstract available. PMID 35595723
- [Background] Bachert C, Zhang N, Holtappels G, De Lobel L, van Cauwenberge P, Liu S, Lin P, Bousquet J, Van Steen K. Presence of IL-5 protein and IgE antibodies to staphylococcal enterotoxins in nasal polyps is associated with comorbid asthma. J Allergy Clin Immunol. 2010 Nov;126(5):962-8, 968.e1-6. doi: 10.1016/j.jaci.2010.07.007. PMID 20810157
- [Background] Han JK, Bachert C, Fokkens W, Desrosiers M, Wagenmann M, Lee SE, Smith SG, Martin N, Mayer B, Yancey SW, Sousa AR, Chan R, Hopkins C; SYNAPSE study investigators. Mepolizumab for chronic rhinosinusitis with nasal polyps (SYNAPSE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 Oct;9(10):1141-1153. doi: 10.1016/S2213-2600(21)00097-7. Epub 2021 Apr 16. PMID 33872587
- [Background] Howarth P, Chupp G, Nelsen LM, Bradford ES, Bratton DJ, Smith SG, Albers FC, Brusselle G, Bachert C. Severe eosinophilic asthma with nasal polyposis: A phenotype for improved sinonasal and asthma outcomes with mepolizumab therapy. J Allergy Clin Immunol. 2020 Jun;145(6):1713-1715. doi: 10.1016/j.jaci.2020.02.002. Epub 2020 Feb 19. No abstract available. PMID 32084443
- [Background] Detoraki A, Tremante E, D'Amato M, Calabrese C, Casella C, Maniscalco M, Poto R, Brancaccio R, Boccia M, Martino M, Imperatore C, Spadaro G. Mepolizumab improves sino-nasal symptoms and asthma control in severe eosinophilic asthma patients with chronic rhinosinusitis and nasal polyps: a 12-month real-life study. Ther Adv Respir Dis. 2021 Jan-Dec;15:17534666211009398. doi: 10.1177/17534666211009398. PMID 33910399
- [Background] Dima E, Kyriakoudi A, Kaponi M, Vasileiadis I, Stamou P, Koutsoukou A, Koulouris NG, Rovina N. The lung microbiome dynamics between stability and exacerbation in chronic obstructive pulmonary disease (COPD): Current perspectives. Respir Med. 2019 Oct;157:1-6. doi: 10.1016/j.rmed.2019.08.012. Epub 2019 Aug 21. PMID 31450162
- [Background] Logotheti M, Agioutantis P, Katsaounou P, Loutrari H. Microbiome Research and Multi-Omics Integration for Personalized Medicine in Asthma. J Pers Med. 2021 Dec 5;11(12):1299. doi: 10.3390/jpm11121299. PMID 34945771
- [Background] Agioutantis PC, Loutrari H, Kolisis FN. Computational Analysis of Transcriptomic and Proteomic Data for Deciphering Molecular Heterogeneity and Drug Responsiveness in Model Human Hepatocellular Carcinoma Cell Lines. Genes (Basel). 2020 Jun 5;11(6):623. doi: 10.3390/genes11060623. PMID 32517019
- [Background] Agioutantis PC, Kotsikoris V, Kolisis FN, Loutrari H. RNA-seq data analysis of stimulated hepatocellular carcinoma cells treated with epigallocatechin gallate and fisetin reveals target genes and action mechanisms. Comput Struct Biotechnol J. 2020 Mar 18;18:686-695. doi: 10.1016/j.csbj.2020.03.006. eCollection 2020. PMID 32257052
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Background] Chan R, RuiWen Kuo C, Lipworth B. Real-life small airway outcomes in severe asthma patients receiving biologic therapies. J Allergy Clin Immunol Pract. 2021 Jul;9(7):2907-2909. doi: 10.1016/j.jaip.2021.01.029. Epub 2021 Feb 2. No abstract available. PMID 33545398
- [Background] Graff S, Brusselle G, Hanon S, Sohy C, Dupont L, Peche R, Michils A, Pilette C, Joos G, Lahousse L, Lapperre T, Louis R, Schleich F. Anti-Interleukin-5 Therapy Is Associated with Attenuated Lung Function Decline in Severe Eosinophilic Asthma Patients From the Belgian Severe Asthma Registry. J Allergy Clin Immunol Pract. 2022 Feb;10(2):467-477. doi: 10.1016/j.jaip.2021.09.023. Epub 2021 Sep 23. PMID 34563736
- [Background] McMurdie PJ, Holmes S. phyloseq: an R package for reproducible interactive analysis and graphics of microbiome census data. PLoS One. 2013 Apr 22;8(4):e61217. doi: 10.1371/journal.pone.0061217. Print 2013. PMID 23630581
- [Background] Bagci C, Beier S, Gorska A, Huson DH. Introduction to the Analysis of Environmental Sequences: Metagenomics with MEGAN. Methods Mol Biol. 2019;1910:591-604. doi: 10.1007/978-1-4939-9074-0_19. PMID 31278678